CLINICAL TRIAL: NCT00838942
Title: Cataract Surgery Benefice in Improvement of Behaviour, Autonomy and Mood for Alzheimer Patients.
Brief Title: Life From Vision in Alzheimer Disease
Acronym: VIVA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P 010110
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-06

CONDITIONS: Alzheimer Disease; Cataract
Keywords: Eyes disease and dementia.; Cataract surgery in the patient with dementia.; Visual hallucinations; Visual acuity,; Specific eye pathologies in Alzheimer's disease.; Improvement of behaviour,; Improvement of autonomy; Improvement of mood; Cataract extraction in Alzheimer disease patient
MeSH Terms: conditions — Alzheimer Disease; Cataract; Dementia; Hallucinations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients suffering from both Alzheimer's disease and low vision due to a bilateral impeding cataract.
  Interventions: Behavioral: Questionaries

INTERVENTIONS:
Behavioral: Questionaries — MMS (Mini Mental Status), ADAS-cog Alzheimer Disease Assessment Scale for cognitive functions, NPI (Neuropsychiatric Inventory) for behavior troubles, IADL (Instrumental Activities of Daily) for autonomy evaluation, GDS (Geriatric Depression Scale) or Cornell Scale (Cornell Scale for Depression in Dementia) for mood troubles.

SUMMARY:
The VIVA study is focused on Alzheimer's disease patients with a low vision due to a bilateral cataract. The aim is to study cataract surgery results on patients' autonomy, behaviour, and mood. In fact those dement elderly patients suffer from a progressive loss of superior functions, with loss of autonomy, behaviour and mood degradation, associated with physical disabilities. The work hypothesis is that a loss of sensorial functions, particularly visual, is an aggravating factor of NEURO-cognitive troubles and absence of communication with outside circle. The protocol consists in investigating superior functions, autonomy, and behaviour troubles of the participating patients, with the help of a series of neuropsychological tests used one month before and three months after cataract operation on the eye with the worst vision. Independently of the study, patients must have given an informed consent to cataract surgery. Their participation lasts 4 months+/- 1 month. The aim of the study is to evaluate whether the cataract surgery improves patients' behaviour, autonomy and mood and possibly to show evidence onf drawbacks in of such a practice.The main objective targets to cataract surgery benefice on patients suffering from both Alzheimer's disease and impeding cataract, aiming to improve behaviour troubles. The specific objective is to measure this benefice in correlation with visual acuity improvement.

DETAILED DESCRIPTION:
VIVA study aims to evaluate cataract surgery results on Alzheimer patients regarding behavior, autonomy and mood. Patients studied are elderly people suffering from both Alzheimer's disease and low vision due to a bilateral impeding cataract. Designed patients come from Ile-de-France-area geriatrics departments.

Methods: the trial consists in a series of neuropsychological tests involving both subject of the study and a close parent one-month before and three months after surgery of the most affected eye. Each patient is under investigation during 4+/1 months. The tests used are the MMS (Mini Mental Status), ADAS-cog Alzheimer Disease Assessment Scale for cognitive functions, NPI (Neuropsychiatric Inventory) for behavior troubles, IADL (Instrumental Activities of Daily) for autonomy evaluation, GDS (Geriatric Depression Scale) or Cornell Scale (Cornell Scale for Depression in Dementia) for mood troubles. All data are registered along as well as medical treatments and severe side effects.

Practical method:An ophthalmologic surgery department head operates on the patients at National Ophthalmologic Hospital "QUINZE VINGT" in Paris.The surgery involves the eye with the worst vision. Study analysis does not take into account the results of the second eye intervention. The surgery consists in a phacoemulsification and setting of an acrylic implant in the posterior chamber. Patients care consists in the usual procedures. The intervention is performed under regional anesthesia exceptionally general anesthesia. A three-day hospitalization is regular considering patients' fragility.The aim of the study is to analyze 3 months after cataract surgery, the different neuropsychological tests, with the help of appropriate statistics. The main endpoint criterion will be the NPI-test improvement between the one-month test before surgery and the three-month test after. A correlation between visual acuity improvement and NPI-test improvement will be verified. The second endpoint criterion will be the study of other scores (MMS, IADL, ADAS-cog, GDS or Cornell test), in a matched-way. If improvement is noted, a regression logistic study will permit to study improvement predictive factors. Each participant will take part in the study during 4+/-1 months.Study rationale and literature data abstract.Cataract treatment, restoring a better visual function, is greatly beneficial upon life quality of elderly people, as largely demonstrated (1, 2). Several studies, based on cognitive functions, daily life activities, and mood, showed a significant amelioration of elderly people operated on for cataract, in comparison with those who refused the intervention (3). Benefice is less in case of ocular co morbidity or in some very old patients (4).Cataract surgery on elderly patients suffering from cognitive decline has given rise to very few studies. Nevertheless, correlation between low vision and cognitive alteration is well established. In France, a Health High Authority (HHA) report devoted to cataract surgical treatment evaluation, based on literature data and experts opinion, was published in 2000 (6). The report dealt with the taking in care of demented or low mental capacities patients. It regretted that very few trials were undertaken for this problem.. In case of beginning dementia, the experts thought that cataract surgery visual benefice is limited. It seldom improves lecture but allows patients to watch television more and makes contacts with neighbors easier. In case of advanced dementia, the authors thought that surgery would worsen rapidly patients. The report evoked as well the paternalistic decisions taken without any dialogue with the involved patient and raised ethical issues. Still to-day, in case of dementia, the cataract management remains an actual problem. This is a challenge for closes, guardians, geriatrics', ophthalmologists and sometimes the decision is opposed to patients' feelings (8).One of the studies cited in the HHA report, based on few low-vision patients, showed after cataract surgery, a light improvement of mental status, everyday life but poor results on depression. After surgery, patients felt that they were not as fragile as they had thought, that they endured the operation and felt better after (9). In 2003, a Japanese study dealt with cognitive functions of 40 demented patients suffering from cataract. Results and showed that among the 20 patients who chose to be operated on, 60% were improved, 35% were unchanged, and 5% worsened (10). By extensive neuropsychological investigations on Alzheimer' patients, the VIVA study would show the impact of visual function improvement on cognitive functions, psychological and behavioural troubles, autonomy, and mood perturbations. Pointing out the objectives upon improvement of neuropsychiatric survey, namely the NPI test, the study would permit to precise the low-vision cataract role on patients' comportment troubles which are a cause of burn-out for caring people. It is clearly demonstrated that delirious manifestations, notably visual hallucinations are frequent in demented persons and in patients with low vision as well (9). In low-vision patients, it seems that only the cataract is significantly linked to visual hallucinations (10). The VIVA study aims to show also the benefice of a better visual function on behavioural non-disturbing troubles such as apathy and inhibition. Therefore, we would like to stress the cataract management benefits on Alzheimer's disease patients. Particularly, we intend to precise the extent of expected patients' improvement and to measure the correlation with visual acuity improvement

ELIGIBILITY:
Inclusion Criteria:

* Signed informed patient's or representative consent for the study
* Patients over 50 years old
* Patients whose bilateral visual acuity is less than 5/10, requiring cataract surgery
* Patients suffering from Alzheimer's disease whose MMS score test is between 10 and 25 (10<MMS≤25)

Exclusion Criteria:

* Patient's or representative's refusal
* NEURO-ocular disease resulting in a severe vision impairment
* Severe and evolving disease involving vital prognosis at short term

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients studied are elderly people suffering from both Alzheimer's disease and low vision due to a bilateral impeding cataract
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2004-12; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Improvement score of the NPI (Neuropsychiatric Inventory). The improvement is based on the increase by 1 point on the score of NPI | 3 month after cataract surgery

SECONDARY OUTCOMES:
Improvement score of MMS(Mini mental status), of ADAS-COG(Alzheimer disease Assessment scale for cognitive function), IADL(Instrumental activity on daily) and GDS(Geriatric depression scale). | 3 month after cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte GIRARD, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Tenon, Service Ophtalmologie, Paris, France